

| Official Title: | Impact of Visual Arts Immersion on Cultural Competency and Self-<br>reflection Among Nurses Working in an Academic Health System |
|---|---|
| NCT Number: | NCT05877976 |
| Study Number: | 23-00530 |
| Document Type: | Informed Consent Form |
| Date of the Document: | • June 19, 2023 |

# **Key Info and Consent Form**

| Record ID |
|-----------|

Title of Study:

Impact of visual arts immersion on cultural competency and self-reflection among nurses working in an academic health system s23-00530

Principal Investigator:

Lita Anglin NYU Health Sciences Library NYU Langone Health 577 First Avenue, New York, NY 10016 Lita.Anglin@nyulangone.org (212) 263-2519

**Emergency Contact:** 

Lita Anglin Lita.Anglin@nyulangone.org (212) 263-2519

Key Study Information Form

You are being invited to take part in a research study. Your participation is voluntary which means you can choose whether or not you want to take part in this study.

### Purpose of the Research Study

The purpose of this study is to explore the impact of a structured art immersion program on perceived cultural competence and self-reflective skills in nurses working in an academic health system. We are asking you to take part in this research study because you are a registered nurse employed at NYU Langone Health.

### Other Key Information

Participation in this study will involve attending 2 art workshops and completing several surveys over a 6-month period. The first workshop will take place at the Metropolitan Museum of Art (MET) and the second workshop will take place virtually over WebEx. Each workshop will be 90 minutes. You will be asked to complete surveys before the first workshop and after the second workshop.

### Foreseeable Risk and Benefits

A comprehensive list of all possible risks and discomforts related to this research is included in the full consent. The most common risk is loss of confidentiality. You may or may not benefit personally from being in this study. Information from this study will give us better insight into the structured at immersion program. We hope other people might benefit from this study in the future.

### Alternatives to Participation

You may choose not to participate or withdraw your participation at any time with no consequence. Your decision to participate, not to participate, or withdraw from the study will not affect your employment, salary, or performance evaluation.

For in-depth details regarding this study, please refer to the full informed consent document attached. For questions and concerns regarding any of this information, contact Lita Anglin at Lita.Anglin@nyulangone.org.

projectredcap.org REDCap®

#### **Informed Consent**

1. About volunteering for this research study

You are being invited to take part in a research study. Your participation is voluntary which means you can choose whether or not you want to take part in this study. Your employment, salary, or performance evaluation will not be affected by your decision whether or not to participate in this study. People who agree to take part in research studies are called "subjects" or "research subjects". These words are used throughout this consent form. Before you can make your decision, you will need to know what the study is about, the possible risks and benefits of being in this study, and what you will have to do in this study. You may also decide to discuss this study and form with your family or friends. If you have any questions about the study or about this form, please ask us. If you decide to take part in this study, you must sign this form. We will give you a copy of this form signed by you for you to keep.

2. What is the purpose of this study?

The purpose of this study is to explore the impact that a structured art immersion program has on perceived self-reflective skills and cultural competence in nurses working in an academic health system.

- 3. How long will I be in the study? How many other people will be in the study? Participation in this study will involve attending 2 art workshops and completing several surveys over a 6-month period. Each workshop will be 90 minutes. The estimated time it will take for you to complete the surveys is approximately 30 minutes. We are expecting to have up to 60 registered nurses from across NYULH campuses take part in the study.
- 4. What will I be asked to do in the study? If you choose to take part in the study, we will ask you to sign this consent form first. The following will also take place:

You will be asked to provide your email or cell phone of choice so we may communicate study information, reminders, and surveys via email or text message. You will then be asked to complete a demographic survey, the Interpersonal Reactivity Index (IRI) and the Cultural Assessment Survey (CAS). The demographic survey contains questions about age, race/ethnicity, gender, years of nursing experience, NYULH campus, specialty, shift time, and role (clinical or nurse leader). CAS measures cultural awareness, sensitivity, knowledge and skills. IRI measures four separate aspects of empathy and its relationships with measures of social functioning, self-esteem, emotionality, and sensitivity to others.

Following completion of the surveys you will be asked to sign up for 2 art immersion classes. You will be offered 4 dates to sign up for the art immersion classes. The first class will be an in-person class at the Metropolitan Museum of Art (MET) located on 5th Ave and 86th New York, NY. The second class will be virtual via WebEx. Each class will last 60 minutes. There will also be an optional independent self-directed reflective exercise with art materials and prompts provided by the MET. At 6 months (after your second class) you will be asked to complete the IRI and the CAS surveys again and additionally complete a short qualitative survey about the overall impact of the art immersion program on your work and life. You are free to skip questions you do not want to answer. Any identifiable information (email or cell phone number) collected and/or used for the purposes of this research will not be used or distributed for future research studies.

#### COMMUNICATING WITH THE RESEARCH TEAM VIA TEXT MESSAGE

Researchers may be need to communicate with you about information relevant to this research study. The Research Team will usually contact you for these purposes by phone, but if you have given the Researchers your email address and mobile/cell phone number and permission to send a text message, the Research Team may contact you that way. When the Research Team sends email messages that include identifiable health information, they will use encrypted messaging (e.g. SendSafe). When the Research Team uses texting over mobile/cell phones there is no way to encrypt the message. This means that information you send or receive by text message is unencrypted and could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier. Therefore, text messages carry security and privacy risks.

Below are some important points about texting in this research study:

Text messages are not encrypted, and therefore are unsecure and may result in a breach of your confidentiality. You will be responsible for all fees charged by your carrier's service plan for text messaging. This research study and NYU Langone Health will not cover the cost related to any increased charges, data usage against plan limits or changes to data fees from research texts. Text messages will only be read during regular business hours. However, if you have a scheduled study visit outside of business hours, you may receive a text in relation to this visit outside of regular business hours. Text messaging should not be used in case of an emergency. If you experience a medical emergency, call 911 or go to the nearest hospital emergency department. You may decide to not send or receive text messages with the research staff associated with this research study at any time. You can do this in person or by sending the Research Team a text message that says "Stop Research Text." Your agreement applies to this research study only. Agreeing to other texts from NYU Langone Health, for example appointment reminders, is a separate process. Opting out of other texts from NYU Langone Health is a separate process as well. Please make sure to keep the Research Team updated if your mobile/cell phone number changes during the study.

\*\*Projectredcap.org\*\*

\*\*Projectredcap.org\*\*

Do you agree to receive texts from this research group?

This is not a requirememnt of participation. You will have an oppoturnity to select your communication preferences (text or email) at the end of this document.

| ○ Yes, I a | agree to receive | texts from | this research |
|------------|------------------|------------|---------------|
| aroup | | | |

 No, I do not agree to receive texts from this research group

## **Informed Consent, continued**



06/02/2023 2:32pm projectredcap.org

### 5. What are the possible risks or discomforts?

### Risk of Loss of Privacy (Confidentiality)

There is a small risk that people may get to see your information who are not supposed to. We will make sure that the information is collected and placed in REDCap and your name will not be collected. Once the study is complete, your email or cell phone number will be destroyed. All de-identified data will be analyzed and reported in aggregate to decrease the chance of being identified. Also, your research data will not be accessible to your supervisors or others who are not directly involved in the research.

### Risk of Completing Survey

Completing surveys may cause discomfort or frustration. You do not have to answer any questions that you do not want to answer, and you are free to withdraw from this study at any time. Risk of Communicating with Research Team via Text Message In this study you may receive texting over mobile/cell phones and this method of communication may result in a breach of your confidential information because text messages to mobile/cell phones are not encrypted. This means that information you send or receive by text message could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier.

#### Other Risks

Another risk is the inconvenience from committing to attending two art classes.

#### 6. What if new information becomes available?

During the course of this study, we may find more information that could be important to you. This includes information that might cause you to change your mind about being in the study. We will notify you as soon as possible if such information becomes available.

### 7. What are the possible benefits of the study?

You may or may not develop increased self-reflective skills that benefit your performance and awareness of connections in nursing practice. The results of this study will help to guide future interventions to assist nurses in developing self-reflective and cultural competency skills that translate to the workplace setting.

### 8. What other choices do I have if I do not participate?

You do not need to participate in this study, it is completely voluntary. Your decision to participate, not to participate, or withdraw from the study will not affect your employment, salary, or performance evaluation.

### 9. Will I be paid for being in this study?

You will not be paid for participating in this study. You will be provided with a travel stipend of \$50, complimentary entry to the museum to participate in the class, plus an additional complimentary ticket to be used at any other time that you wish. You will also be provided with a bag of art supplies that are yours to keep.

### 10. Will I have to pay for anything?

You will have to initially pay for your own transportation to and from The MET and you will be provided a \$50 gift card to use to cover that expense.

#### 11. What happens if I am injured from being in the study?

For medical emergencies contact 911. If you think you have been injured as a result of taking part in this research study, tell the principal investigator as soon as possible. The principal investigator's name and phone number are listed at the top of page 1 of this consent form. We will offer you the care needed to treat injuries directly resulting from taking part in this research. There are no plans for NYU Langone Health to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

### 12. When is the study over? Can I leave the study before it ends?

This study is expected to end after all participants have completed all the surveys, and all information has been collected at the 6-month mark. This study may also be stopped, or your participation ended at any time by the study team without your consent because:

The principal investigator feels it is necessary for your safety. Such an action would not require your consent, but you will be informed if such a decision is made and the reason for this decision. You have not followed study instructions. The principal investigator or other body responsible for monitoring the study has decided to stop the study. If you decide to participate, you are free to leave the study at any time. Leaving the study will not affect your employment, salary, or performance evaluation.

### 13. How will you protect my confidentiality?

We are committed to protecting the privacy and confidentiality of your information. Your research data will not be accessible to your supervisors or others who are not directly involved in the research. The risk of being identified as நடிந்து நூர்கள் நடிந்து நூர்கள் மான்ற முறையாக மான்ற முறையாக மான்ற முறையாக மான்ற முறையாக மு

of choice. The researchers will make sure that the information is collected and placed in REDCap and your name will not be collected. Once the study is complete your email and/or phone number will be destroyed. All de-identified data will be analyzed and reported in aggregate to decrease the change of being identified.

What information may be used or shared with others in connection with this study? Your survey responses may be used and shared with those individuals listed in this section.

Who may use and share information in connection with this study? The following individuals may use, share, or receive your information for this research study:

The research team, including the Principal Investigator, study coordinators, and personnel responsible for the support or oversight of the study. Study Sponsor: National Network of the Library of Medicine (NNLM) Division of the National Library of Medicine (NLM) 14. The Institutional Review Board (IRB) and how it protects you The IRB reviews all human research studies - including this study. The IRB follows Federal Government rules and

guidelines designed to protect the rights and welfare of the people taking part in the research studies. The IRB also reviews research to make sure the risks for all studies are as small as possible. The NYU Langone Health IRB Office number is 212-263-4110. The NYU Langone Health IRB is made up of doctors, nurses, non-scientists, and people from the Community. 15. Who can I call with questions, or if I'm concerned about my rights as a research subject? If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigator listed on top of the page 1 of this consent form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the Institutional Review Board (IRB) at 212-263-4110. Do you consent to participating in this study? Yes Selecting yes below means you are agreeing to take  $\bigcirc$  No part in this research study as described to you. This means you have read the consent form, your questions have been answered, and you have decided to volunteer. **Contact information and session registration** How would you like to receive communication from the Text research team? **Email** Both Cell phone number (10 digits, beginning with area code) Email address Please select one in-person workshop session, to take O Date 1 place at The Metropolitan Museum of Art (1000 5th Ave. O Date 2 New York, NY 10028, enter at 81st) O Date 1 Please select one virtual session date, to take place via WebEx O Date 2

Clicking submit below will take you to the demographics and baseline survey. Thank you for your participation!